CLINICAL TRIAL: NCT04114201
Title: Evaluation of Zimmer® Patient Specific Instrumentation vs. Conventional Instrumentation in Total Knee Arthroplasty Procedures: Clinical and Economic Outcomes
Brief Title: Clinical Outcome and OR Resource Use of Total Knee Arthroplasty Using Patient-Specific or Conventional Instrumentation
Acronym: TKA PSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA-PSI
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patients were operated consecutively with conventional and patient-specific Instrumentation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSI (Experimental): Patients received TKA using patient-specific Instrumentation.
  Interventions: Procedure: PSI
- Conventional (Active Comparator): Patients received TKA conventional Instrumentation.
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: PSI — Implantation of a Total Knee Arthroplasty patient-specific instrumentation using Zimmer® NexGen Solutions (Zimmer Biomet, Warsaw, IN).
  Arms: PSI
Procedure: Conventional — Implantation of a Total Knee Arthroplasty with conventional using Zimmer® NexGen Solutions (Zimmer Biomet, Warsaw, IN).
  Arms: Conventional

SUMMARY:
Compare OR resource use and clinical Outcome after Total Knee Arthroplasty using Patient-specific or conventional Instrumentation.

DETAILED DESCRIPTION:
The aim of this study was to compare OR resource use and clinical Outcome after Total Knee Arthroplasty (TKA) using Patient-specific (PSI) or conventional Instrumentation.

For this purpose, economic variables of the surgery (number of instrument trays, setup and cut-sew-time), radiological alignment and patient reported outcomes (VAS Pain Scale, Oxford Knee Score, EQ-5D) were assessed. Cost per QALY (quality-adjusted life year) was assessed using the German DRG reimbursement and the EQ-5D.

A total of 139 TKA with PSI or conventional instrumentation were included in three Centers and were assessed before surgery, as well as 6 weeks, 6 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Painful, disabled knee joint resulting from osteoarthritis requiring primary TKA
* Informed Consent: Patient has signed a "Patient Informed Consent.
* Able and willing to undergo a preoperative MRI scan (for PSI cases) and full-leg, standing radiographs (all cases)
* Able and willing to follow instructions and complete follow-up
* Patient receiving Zimmer NexGen Solutions CR-Flex (including Gender Solutions)

Exclusion Criteria:

* Patient is skeletally immature
* Active Infection (including septic knee, distant infection, or osteomyelitis)
* Severe hip arthrosis
* Neurological disorders (including, but not limited to Parkinson's disease)
* Prior unicompartmental knee arthroplasty, TKA, knee fusion or patellectomy
* Hip or knee ankylosis
* Either rheumatoid or post-traumatic knee arthritis
* Scheduled for simultaneous bilateral TKA
* Indications of intra- and/or extra-articular deformations that would inhibit the use of PSI guides
* Any metal within 150 mm of the joint line for the operative-side knee
* Knee deformities greater than 15 degrees of fixed varus, valgus, or flexion contracture on initial physical examination
* An existing condition that would, in the opinion of the investigator, compromise participation or follow-up in this study
* A female who is pregnant or lactating
* Current involvement in any personal injury litigation, medical-legal or worker's compensation claims
* Arterial disease or stents that would exclude the use of a tourniquet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-08-02 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
OR time | during surgery
  Operating Room (OR) time: incision to Close in minutes

SECONDARY OUTCOMES:
OR resource use: number of instrument trays | during surgery
  OR Efficiency measured by number of instrument trays used
OR Setup Time | during surgery
  Operating Room (OR) Setup Time in minutes
Oxford Knee Score | 1 year after surgery
  clinical outcome measured by the Oxford Knee Scoring System. The Oxford Knee Score is aggregated to a single score where 0 is the worst and 48 is the best Outcome.
visual analog scale (VAS) | 1 year after surgery
  patient-reported pain scores as measured by the visual analog scale (VAS), ranging from 0 (worst) to 10 (best).
device alignment | 1 year after surgery
  device alignment as determined using radiographs (A/P long-standing and lateral films)
EQ-5D-3L | 1 year after surgery
  patients' health-related Quality of life is measured by the EQ-5D-3L, which aggregates to a single index where 0 is the worst and 1 is the best outcome

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Department for Orthopaedic and Trauma Surgery, Schön Klinik Lorsch, Lorsch, Hesse
  - Department for Orthopaedic and Trauma Surgery, Helios Kliniken Mittelweser, Nienburg, Lower Saxony
  - University Center of Orthopaedics and Traumatology, University Medicine Carl Gustav Carus Dresden, TU Dresden, Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No